CLINICAL TRIAL: NCT06027437
Title: A Phase 1, Open-label, Randomized, Single-dose, 3-Period, 3-Sequence Crossover Study to Assess the Relative Bioavailability of the Intended Commercial Formulation Versus the Previous MyoKardia Formulation of Danicamtiv and to Assess the Effect of Food on the Pharmacokinetics of the Intended Commercial Formulation in Healthy Adult Participants
Brief Title: A Study to Assess the Relative Biological Availability and the Effect of Food on the Drug Levels of Danicamtiv in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CV028-1012
Record Dates: First submitted 2023-08-31; First posted 2023-09-07 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Healthy Volunteers
Keywords: BMS-986434; MYK-491; Healthy; Biological Availability; Food Effect

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment A (Experimental)
  Interventions: Drug: Danicamtiv
- Treatment B (Experimental)
  Interventions: Drug: Danicamtiv
- Treatment C (Experimental)
  Interventions: Drug: Danicamtiv

INTERVENTIONS:
Drug: Danicamtiv — Specified dose on specified days.
  Other Names: BMS-986434; MYK-491

SUMMARY:
The purpose of this study is to assess the relative biological availability and the effect of food on the drug levels of Danicamtiv in health adults.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) of 18.0 kg/m2 to 30.0 kg/m2 inclusive
* Participants with resting heart rate ≥ 55 bpm
* Seasonal allergies that do not require medication at the time of the study are acceptable

Exclusion Criteria:

* Any acute or chronic medical illness
* Head injury, intracranial tumor, or aneurysm within 2 years prior to screening
* History of chronic gastrointestinal disorders or gastrointestinal (GI) surgery (including cholecystectomy) that could impact on drug and food absorption and/or drug excretion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to day 16
Area under the plasma concentration time curve from time zero extrapolated to infinite time (AUC(INF)) | Up to day 16
Area under the plasma concentration time curve from time zero to the time of the last quantifiable concentration (AUC(0-T)) | Up to day 16

SECONDARY OUTCOMES:
Time of maximum observed plasma concentration (Tmax) | Up to day 16
Terminal elimination half-life (T-HALF) | Up to day 16
Apparent total body clearance (CLT/F) | Up to day 16
Apparent volume of distribution (Vz/F) | Up to day 16
Number of participants with Adverse Events (AEs) | Up to day 43
Number of participants with Serious Adverse Events (SAEs) | Up to day 43
Number of participants with vital sign abnormalities | Up to day 16
Number of participants with Electrocardiogram (ECG) abnormalities | Up to day 16
Number of participants with Physical Examination (PE) abnormalities | Up to day 16
Number of participants with clinical laboratory abnormalities | Up to day 16

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Anaheim Clinical Trials, Anaheim, California, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSStudyConnect.com